CLINICAL TRIAL: NCT04991129
Title: A Dose Escalation and Dose Expansion Study of WJ01024 to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy for Patients With Advanced Cancer
Brief Title: The Safety and Efficacy of Multiple-dose of WJ01024 in Subject With Advanced Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Due to a change in the development strategy, the sponsor decided to terminate the study on May 28, 2025
Sponsor: Suzhou Junjing BioSciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JJSW-01
Record Dates: First submitted 2021-07-14; First posted 2021-08-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Advanced Hematologic Malignancies; Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Sequential
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (10):
- WJ01024 5mg QD repeat dose every 28 days (Experimental)
  Interventions: Drug: WJ01024
- WJ01024 5mg BID repeat dose every 28 days (Experimental)
  Interventions: Drug: WJ01024
- WJ01024 10mg BID repeat dose every 28 days (Experimental)
  Interventions: Drug: WJ01024
- WJ01024 40mg BIW repeat dose every 28 days (Experimental)
  Interventions: Drug: WJ01024
- WJ01024 60mg BIW repeat dose every 28 days (Experimental)
  Interventions: Drug: WJ01024
- WJ01024 80mg BIW repeat dose every 28 days (Experimental)
  Interventions: Drug: WJ01024
- WJ01024 60mg QW repeat dose every 28 days (Experimental)
  Interventions: Drug: WJ01024
- WJ01024 80mg QW repeat dose every 28 days (Experimental)
  Interventions: Drug: WJ01024
- WJ01024 50mg QW repeat dose every 28 days (Experimental)
  Interventions: Drug: WJ01024
- WJ01024 40mg QW repeat dose every 28 days (Experimental)
  Interventions: Drug: WJ01024

INTERVENTIONS:
Drug: WJ01024 — 5mg QD: WJ01024, Q4W, once per day
  Arms: WJ01024 5mg QD repeat dose every 28 days
Drug: WJ01024 — 5mg BID: WJ01024, Q4W, twice per day
  Arms: WJ01024 5mg BID repeat dose every 28 days
Drug: WJ01024 — 10mg BID: WJ01024, Q4W, twice per day
  Arms: WJ01024 10mg BID repeat dose every 28 days
Drug: WJ01024 — 40mg BIW: WJ01024, Q4W, twice per week
  Arms: WJ01024 40mg BIW repeat dose every 28 days
Drug: WJ01024 — 60mg BIW: WJ01024, Q4W, twice per week
  Arms: WJ01024 60mg BIW repeat dose every 28 days
Drug: WJ01024 — 80mg BIW: WJ01024, Q4W, twice per week
  Arms: WJ01024 80mg BIW repeat dose every 28 days
Drug: WJ01024 — 60mg QW: WJ01024, Q4W, once per week
  Arms: WJ01024 60mg QW repeat dose every 28 days
Drug: WJ01024 — 80mg QW: WJ01024, Q4W, once per week
  Arms: WJ01024 80mg QW repeat dose every 28 days
Drug: WJ01024 — 50mg QW: WJ01024, Q4W, once per week
  Arms: WJ01024 50mg QW repeat dose every 28 days
Drug: WJ01024 — 40mg QW: WJ01024, Q4W, once per week
  Arms: WJ01024 40mg QW repeat dose every 28 days

SUMMARY:
A clinical study of WJ01024 in subjects with advanced cancer in China, to evaluate the safety, tolerability, PK and efficacy of WJ01024. This study includes a dose escalation part and a dose expansion part. Patients receive WJ01024 on Day 1 and Day 3 of each week, 4 weeks as a cycle, until disease progression, or intolerable toxicity , withdrawal of consent, or end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion criteria：

1. Patients with advanced malignant neoplasms definitively diagnosed by pathology and/or cytology who have failed to respond to conventional treatment or are lacking effective treatment;
2. For patients with solid tumors, there should be evaluable or measurable tumor lesions according to RECIST 1.1 criteria (not for dose-climbing phase);
3. Males and females ≥ 18 and ≤ 75 years of age,ECOG performance status of 0~1;
4. Life expectancy ≥3 months;
5. The functions of the major organs were basically normal, and the following laboratory tests were performed within 7 days before the first administration of the study drug (no blood transfusion or colony-stimulating factor was administered within 14 days before the examination);
6. For premenopausal women who are likely to have children, a pregnancy test must be performed within 7 days before the first use of the study drug. The blood pregnancy test must be negative and must be non-lactating.All enrolled patients (both male and female) should take adequate barrier contraception throughout the treatment period and 3 months after the end of treatment;
7. Voluntary participant in this drug clinical trial, able to understand and sign the informed consent.

Exclusion criteria

1.Pregnant or lactating women; 2.Suffer from other serious complications (such as uncontrolled infection, myocardial infarction within 6 months, uncontrolled hypertension and thromboembolic disease); 3.There was active graft rejection at the time of enrollment (after allogeneic stem cell transplantation); 4.Who is not suitable for the study after laboratory examination (blood routine, urine routine, blood biochemical, blood coagulation function) or as judged by the study physician; 5.≥ Grade 2 toxicity after previous treatment;6.Patients with grade 2 or more neuropathy; 7.A person suffering from an uncontrollable mental illness; 8.Have a history of drug abuse or urine drug screening positive; 9.Heart disease: New York heart association (NYHA) > class II congestive heart failure, unstable angina (resting angina symptoms), new angina (within 6 months before entering the study), into the group of the first six months of myocardial infarction, or need anti-arrhythmic treatment for arrhythmia (allows the use of beta blockers, calcium channel blockers and digoxin); 10.Alcoholics or those who consume more than 28 units of alcohol per week (1 unit = 285 mL beer or 25 mL spirits (40%v/v) or 1 glass [100ml] of wine); 11.Patients with active hepatitis B, hepatitis C, HIV (+) and syphilis antibody (+);Patients with HBsAg or core antibody (HBcAb) positivity need to be tested for HBV-DNA, and HBV-DNA is lower than the upper limit of normal to be enrolled.Patients with hepatitis C virus antibody (HCV Ab) positive should be tested for HCV RNA, and those below the upper limit of normal can be enrolled.

12.Requiring long-term corticosteroids or other immunosuppressive therapy, such as those who have had organ transplants; 13.Other conditions considered ineligible by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2025-05-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
The incidence of adverse events (AE) and serious adverse events (SAE) were assessed | 2 years
  Incidence and severity of adverse events (AE) and serious adverse events (SAE) as assessed according to NCI-CTCAE 5.0, as well as abnormalities in vital signs, electrocardiogram, and laboratory tests

SECONDARY OUTCOMES:
ORR | 2 years
  DLT, MTD, RP2D, Number of participants and severity with treatment-related Adverse events as assessed by CTCAE V5.0
DOR | 2 years
  Duration of Response
DCR | 2 years
  Disease Control Rate
PFS | 2 years
  Progression-free survival
Cmax | 2 years
  Maximum Plasma Concentration
Tmax | 2 years
  Time to Cmax
AUC0-t | 2 years
  Area under the concentration versus time curve from time 0 to the last measurable concentration
AUC0-inf | 2 years
  AUC from time 0 to infinity
Kel | 2 years
  Elimination rate constant
t1/2 | 2 years
  Elimination half life time
CL/F | 2 years
  Clearance
Vd/F | 2 years
  Apparent volume of distribution
Rac | 2 years
  Accumulation factor

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (4):
- China (4):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Harbin The First Hospitall, Harbin, Heilongjiang
  - Jilin Cancer Hospital, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: No